

January 25, 2019

Martha Kruhm, MS RAC
Head, Protocol and Information Office
Quality Assurance Section
CTEP, DCT, NCI
6130 Executive Blvd, EPN Room 7000
Bethesda, MD 20892

Dear Dr. John J. Wright:

Enclosed is Addendum #18 to EAY131-G, Molecular Analysis for Therapy Choice (MATCH): MATCH Treatment Subprotocol F: Phase II Study of Crizotinib in Patients with ROS1 Translocations (Other Than Patients with Non-Small Cell Lung Cancer).

This addendum is in response to Dr. John J. Wright's January 22, 2019 Request for Rapid Amendment for Crizotinib.

The following revisions to EAY131-G protocol have been made in this addendum:

| | Section | Change |
|---|---|---|
| 1. | Cover Page | Updated Version Date. |
| 2. | 3.3 | Updated the Crizotinib CAEPR list with Version 2.3, October 30, 2018. |

The following revisions to EAY131-G Informed Consent Document have been made in this addendum:

| | Section | Change |
|---|---|---|
| 1. | Page 1 | odated Version Date. |
| 2. | What possible risks can I expect from taking part in this study? | Updated the Crizotinib risk list with Version Date October 30, 2018. |

If you have any questions regarding this addendum, please contact <a href="mailto:aagu@ecog-acrin.org">aagu@ecog-acrin.org</a> or 857-504-2900.

We request review and approval of this addendum to EAY131-G so ECOG-ACRIN may activate it promptly.

Thank you.

#### Sincerely,

#### Pamela Cogliano

#### Senior Director of Protocol Development

#### **Enclosure**

CC: David S. Hong, MD Anna F. Farago, MD, PhD

Alice Chen, MD

Keith Thomas Flaherty, MD Barbara A. Conley, MD Peter O'Dwyer, MD Mickey Williams, PhD Stanley Hamilton, MD Lisa McShane, PhD Larry Rubinstein, PhD Robert Gray, PhD Shuli Li, PhD

Lalitha Shankar, MD, PhD Susanna Lee, MD, PhD

Constantine Gastonis, PhD Paolo Caimi, MD Shaji Kumar, MD Carlos Arteaga, MD

Edith Mitchell, MD John J. Wright, MD

Angela Chen Daniel Reeve Lyndsay Harris, MD James Tricoli, PhD

Bruce Giantonio, MD Donna Marinucci

Kerry Higgins Gayle Ipock

Jean MacDonald Carol Chami, RN Julianne Human

Kelly Redmond Becky Fillingham Jeffrey Zhang

Kevin Pollard Amy Li

Abuchi Agu Michael T. Balco Lauren Lambert Cayden Maican

Margaret Cavenagh

Ben Kim

Alexandra Sachs Russell McDaniel Jennifer VanCamp



# Molecular Analysis for Therapy Choice (MATCH)

# MATCH Treatment Subprotocol G: Phase II Study of Crizotinib in Patients with ROS1 Translocations (Other Than Patients with Non-Small Cell Lung Cancer)

TREATMENT SUBPROTOCOL CHAIR: Aaron Mansfield, MD
TREATMENT SUBPROTOCOL CO-CHAIR: Christopher Lieu, MD
TRANSLATIONAL CHAIR: Patrick Forde, MD, MBBCh

Version Date: January 25, 2019 NCI Update Date: August 12, 2015

Rev. 8/15 NOTE: This subprotocol (EAY131-G) should

be used in conjunction with the MATCH Master Protocol (EAY131).

Rev. Add13 NOTE: As of 11/17, all protocol changes will

be noted by addendum number.
please reference the activation memo
for the addendum activation date.

SUBPROTOCOL ACTIVATION DATE

August 12, 2015

SUBPROTOCOL PRE-ACTIVATION DATE

May 29, 2015

Update #1 – Incorporated Prior to Activation

Addendum #1 - 8/15

Update #2 - 8/15

Addendum #2 - 2/16

Addendum #3 – 5/16 Addendum #5 – 12/16

Addendum #7 – 3/17

Addendum #11 - 8/17

Addendum #13

Addendum #18

| Agent | IND# | NSC# | Supply |
|------------|------|--------|--------------|
| Crizotinib | | 749005 | NCI Supplied |

### **Table of Contents**

| Molecular Analysis for Therapy Choice (MATCH) | <u>i</u> |
|---|---|
| MATCH Treatment Subprotocol G: Phase II Study of Crizotinib in Patients with | i |
| ROS1 Translocations (Other Than Patients with Non-Small Cell Lung Cance | r) <u>1</u> |
| Table of Contents | 2 |
| Schema | 4 |
| 1. Introduction | 5 |
| 1.1 Crizotinib | 5 |
| 1.2 Supporting Preliminary Data | <u>7</u> |
| 2. Selection of Patients | <u>9</u> |
| 2.1 Eligibility Criteria | <u>9</u> |
| 3. Criztonib Treatment Plan | 11 |
| 3.1 Administration Schedule | 11 |
| 3.2 Adverse Event Reporting Requirements | <u>11</u> |
| 3.3 Comprehensive Adverse Events and Potential Risks List (CAEPR) for | |
| <u>Crizotinib (PF-02341066, NSC 749005)</u> | |
| 3.4 Dose Modifications | |
| 3.5 Supportive Care | |
| 3.6 Duration of Agent-specific treatment | |
| 3.7 Duration of Follow-Up | |
| 4. Study Parameters. | |
| 4.1 Therapeutic Parameters for Crizotinib Treatment | |
| 5. Drug Formulation and Procurement | |
| 5.1 Crizotinib (NSC #749005) | |
| 6. Translational Studies | |
| 7. References | <u>29</u> |
| Appendix I Pill Calendar | 31 |
| Appendix II CYP3A4 Inducers and Inhibitors | 3 <u>3</u> |
| Appendix III Information On Possible Drug Interactions | 34 |
| Appendix IV Actionable Mutations for Sub-Protocol EAY131-G | 37 |
| Appendix V Medications That May Cause QTc Prolongation | 39 |

#### TREATMENT SUBPROTOCOL CHAIR

Aaron Mansfield, MD Mayo Clinic 200 First St SW Rochester, MN 55905 Phone: 507 293-0569

Fax: 507 284-1803

E-mail: mansfield.aaron@mayo.edu

#### TREATMENT SUBPROTOCOL CO-CHAIR

Christopher Lieu, MD 12801 E. 17<sup>th</sup> Ave, MS 8117 Aurora, CO 80045 Phone: 303-724-6390 Fax: 303-724-3889

E-mail: christopher.lieu@ucdenver.edu

#### TRANSLATIONAL CHAIR

Patrick Forde, MD Johns Hopkins University 1650 Orleans Street, CRB1 Rm G92 Baltimore, MD 21287 Phone: 410-955-3974

Fax: 410-614-9334 E-mail: pforde1@jhmi.edu

### Schema



Cycle = 28 days Accrual Goal: 35

EAY131-G Version Date: January 25, 2019

NCI Update Date: August 12, 2015

#### 1. Introduction

#### 1.1 <u>Crizotinib</u>

Crizotinib is an ATP-competitive small-molecule oral inhibitor of the anaplastic lymphoma kinase, c-MET/hepatocyte growth factor receptor (HGFR), Recepteur d'Origine Nantais (RON), and ROS receptor tyrosine kinases and their oncogenic variants (e.g., c-MET/HGFR mutations and ALK or ROS1 fusion proteins). The rationale for use of this mechanism to treat cancer is supported by an emerging paradigm in oncology that robust clinical efficacy can be obtained with well-tolerated inhibitors directed toward oncogenic tyrosine kinases that are genetically altered through activating mutations, gene translocations, or gene amplification.

#### Clinical Experience with Crizotinib

Crizotinib has been tested in numerous phase I. II and III studies in patients with advanced solid tumors. More than 1511 advanced NSCLC patients have received crizotinib on clinical trials at the dosage of 250mg BID that is approved for advanced ALK-rearranged NSCLC. In the first report of crizotinib for ALKrearranged NSCLC there was an overall response rate of 57% and a 6-month progression free survival of 72% amongst 82 treated patients. An update of this phase 1 trial which included a total of 149 patients reported an overall response rate of 60.8% and a median duration of response of 49.1 weeks.<sup>2</sup> In a separate trial that compared crizotinib in 173 patients to chemotherapy in 174 patients, all with metastatic ALK-rearranged NSCLC, there was a response rate of 65% in the criztonib group compared to 20% in the chemotherapy group. Additionally, median progression free survival was 7.7 months in the crizotinib group compared to 3.0 months in the chemotherapy group.<sup>3</sup> There are few data available on the effects of crizotinib for patients with ROS1-rearranged metastatic NSCLC. The largest study that has been published included 50 patients and demonstrated a 72% response rate and median progression free survival of 19.2 months.<sup>4</sup> ROS1 rearrangements have been identified in other malignancies. There were three patients out of 33 with inflammatory myofibroblastic tumors that harbored a ROS1 rearrangement. The one patient in this study for whom treatment data were available obtained an objective response with crizotinib.5

#### Pharmacokinetics & Metabolism

After a single crizotinib dose of 250 mg, Cmax (peak plasma concentration) was achieved at a median of 4 h, and was associated with a geometric mean terminal half life at steady state of 42 hours. 1-2, 6-7 Age, gender, race, or body weight do not appear to affect crizotinib pharmacokinetics. At the licensed dose of 250 mg BID PO, crizotinib reaches steady state within 15 days. Crizotinib exhibits nonlinear PK with reductions noted in CL/F with multiple dosing compared with single dosing. This may be due to auto-inhibition of CYP3A. Crizotinib PK in ALK-positive NSCLC patients was similar to that seen in patients with other tumor types. The concentration-time profiles and PK parameters of crizotinib in Chinese patients were similar to those observed in Asian (mainly Korean and Japanese) and non-Asian patients.

EAY131-G Version Date: January 25, 2019

NCI Update Date: August 12, 2015

After oral dosing, crizotinib is absorbed with peak plasma concentration occurring between 4-6 hours under fasted condition. The presence of food did not result in clinically meaningful changes in crizotinib PK therefore crizotinib may be taken with or without food.

Crizotinib is highly bound to plasma proteins and is predominantly metabolized by CYP3A. Approximately 53.5% of orally administered crizotinib is excreted unchanged in feces.

#### Safety, Adverse Events and Efficacy of Crizotinib

Crizotinib has primarily been utilized in the setting of patients with ALK rearrangements. In the expanded cohort phase I trial, most subjects tolerated crizotinib well with grade 1 nausea (52%) and diarrhea (46%) being the most common side effects. 1,2 Additionally, 41% of subjects experienced grade 1 visual disturbances most commonly described as trails of light following moving objects. There was one grade 4 elevation in alanine aminotransferase, and one grade 3 episode of pneumonitis. In this trial there was an overall response rate of 57% and a 6-month progression free survival of 72%. Follow up data from this study were reported in 2012 and adverse events are detailed in Table 1. In a phase III study comparing crizotinib to chemotherapy for patients with NSCLC and ALK rearrangements, 172 patients tolerated criztonib relatively well.<sup>3</sup> The most common grade 3 or 4 event was elevated aminotransferase levels (16%). Less common grade 3 or 4 events included nausea (1%), vomiting (1%), constipation (2%), fatigue (2%), dizziness (1%) and dyspnea (4%). The most common adverse events (all grades) were visual disturbances (60%) and diarrhea (60%). In this trial, the patients who received crizotinib had a 65% response rate and a median progression free survival of 7.7 months. Similarly, in a phase I clinical trial for 50 patients with NSCLC and ROS1 rearrangements, crizotinib was well tolerated.<sup>4</sup> There was a similar side effect profile. No grade 4 or 5 events were observed. Grade 3 vomiting or elevated aspartate aminotransferase was seen in one patient each, elevated alanine aminotransferase in two patients, and hypophosphatemia or neutropenia in five patients each. The most common side effect again was grade 1 visual disturbances (82%). There was a 72% response rate and median progression free survival of 19.2 months observed in this clinical trial. Less common adverse events have been described with crizotinib use including hypogonadism and decreased testosterone levels in males.8

| Adverse Events | | | |
|---|---|---|---|
| Study & Population | Selected Adverse Events | All Grades | Grade 3 & 4 |
| | Any Adverse Event | 97% | 24% |
| | Visual Effects | <u>64%</u> | 0% |
| | Nausea | <u>56%</u> | < 1% |
| Kwak et al. NEJM 2010, | Diarrhea | <u>50%</u> | 0% |
| Camidge et.al Lancet Oncol 2012 <sup>1, 2</sup> | Vomiting | <u>39%</u> | < 1% |
| Phase I ALK-rearranged | Peripheral edema | <u>30%</u> | 0% |
| NSCLC | Constipation | <u>28%</u> | < 1% |
| N=149 | Reduced appetite | <u>16%</u> | 0% |
| | Fatigue | <u>16%</u> | 1% |
| | Increased ALT | <u>12%</u> | 4% |
| | Increased AST | <u>10%</u> | 3% |
| | Pnemonitis | <u>&lt; 1%</u> | < 1% |
| Shaw et al. | Visual Effects | 60% | 0% |
| NEJM 2013 <sup>5</sup> | Diarrhea | 60% | 0% |
| Phase III 2 <sup>nd</sup> line ALK- | Nausea | 55% | 1% |
| rearranged NSCLC | Constipation | 42% | 2% |
| N=172 | Elevated ALT/AST | 38% | 16% |

#### 1.2 Supporting Preliminary Data

#### Preclinical Data

Crizotinib has been studied in a variety of in vitro and in vivo model systems to determine potency for inhibition of ALK, c-MET/HGFR, RON, or ROS1 RTK activity, kinase selectivity, antitumor efficacy, PK/PD relationships, and mechanism of action. Crizotinib demonstrated potent concentration-dependent inhibition of the kinase activity of ALK, c-MET/HGFR, RON, and ROS1 in biochemical assays and inhibited phosphorylation and kinase dependent function in cell-based assays. Crizotinib demonstrated potent and selective growth inhibitory activity and induced apoptosis in tumor cells lines exhibiting ALK fusion variants (EML4-ALK) or NPM-ALK), ROS1 fusion variants, or exhibiting amplification of the ALK or c-MET/HGFR gene locus. In vivo, crizotinib demonstrated potent and selective growth inhibitory activity and induced apoptosis in tumor cell lines exhibiting ALK fusion variants (EML4-ALK or NPM-ALK), ROS1 fusion variants, or exhibiting amplification of the ALK or c-MET/HGFR gene locus. In vivo, crizotinib demonstrated antitumor efficacy, including marked cytoreductive antitumor activity, in mice bearing tumor xenografts that expressed ALK fusion variants or activated c-MET/HGFR. The anti-tumor efficacy of crizotinib was dose-dependent and correlated to pharmacodynamic inhibition of phosphorylation of ALK fusion variants (EML4-ALK or NPM-ALK) or c-MET/HGFR in tumors in vivo. The collective rationale for investigation of crizotinib in clinical studies is built on genetic alteration of its molecular targets, its predicted ability to target multiple processes that are common to cancer progression, and preclinical efficacy data.

NCI Update Date: August 12, 2015

#### Rationale for Crizotinib in ROS1-translocated Tumors

Several lines of evidence suggest that ROS1 may represent another therapeutic target of crizotinib. ROS1 encodes a transmembrane protein with an extracellular domain that is partially analogous to fibronectin.<sup>8</sup> Although the function of wild type ROS1 is poorly understood, it is speculated that ROS1 might translate adhesion events to intracellular signaling because of the structural similarities to cell adhesion molecules. The kinase domains of ALK and ROS1 share 77% amino acid identity within the ATP-binding sites, and due to this homology, crizotinib binds with high-affinity to both ALK and ROS1.<sup>8</sup> In cell-based assays for inhibition of autophosphorylation of different kinase targets, both ALK and ROS1 are sensitive to crizotinib, with a half-maximal inhibitory concentration of 40 to 60nM.<sup>8</sup> Preclinical studies have shown that crizotinib potently inhibits ROS1 signaling and cell viability in cell lines expressing ROS1 fusions.<sup>9-12</sup>

The ROS1 proto-oncogene has been identified to be translocated in non-small cell lung cancers and is predicted to exhibit the properties of an "oncogenic driver". In published studies, the frequency of ROS1-positive NSCLC has been examined in 2 studies ranging from 1.7% (18/107) to 2.6% (17/656). 10,13 Patients with adenocarcinoma of lung have demonstrated remarkable responses to crizotinib when their tumor has a ROS1 translocation. An expansion cohort of 50 response-evaluable advanced ROS1-positive NSCLC patients with crizotinib 250 mg BID (NCT00585195) was recently reported, including an ORR of 72% (95% CI: 58–84), with 3 complete responses and 33 partial responses. The median duration of response was 17.6 months (95% CI, 14.5 to not reached), with 25 patients (50%) still in follow-up for progression. Among 30 tumors that were tested, 7 ROS1 fusion partners: 5 known and 2 novel partner genes were identified. The most common ROS1 fusion partner was the gene encoding CD74. Other partner genes included SDC4, EZR, SLC34A2, TPM3, LIMA1, and MSN.

It is anticipated that the frequency of ROS1 translocations across all tumors is relatively rare. However, there have been reports of ROS rearrangements in cancers such as CMML (70%), gastric cancer (5), glioblastoma (incidence unknown), NSCLC (1-2%), cholangiocarcinoma (9%), ovarian cancer (0.5%), colorectal cancer (1%), inflammatory myofibroblastic tumor, angiosarcoma and epithelial hemangioendothelioma. Additional ROS1 fusion partner genes identified in these malignancies included CCDC6, CEP85L, FIG (aka GOPC), KDELR2, KIF5B, LRIG3, TFG, and YWHAE. The dramatic responses and duration of benefit for patients with ROS1 translocations in non-small cell lung cancer argue that, though infrequent, ROS translocations may be a substantial "driver" mutation, and thus, across cancers, and with crizotinib treatment, there may be a response/longer progression-free survival time in any tumor harboring a ROS translocation.

#### 2. Selection of Patients

Each of the criteria in the checklist that follows must be met, along with the eligibility in the main screening study, in order for a patient to be considered eligible for this study. Use the checklist to confirm a patient's eligibility. For each patient, this checklist must be photocopied, completed and maintained in the patient's chart.

In calculating days of tests and measurements, the day a test or measurement is done is considered Day 0. Therefore, if a test is done on a Monday, the Monday four weeks later would be considered Day 28.

ECOG-ACRIN Patient No. \_\_\_\_\_

Patient's Initials (L, F, M)

Physician Signature and Date

| | • | | • | |
|---|---|---|---|---|
| | NOTE: | ;<br>;<br>; | criteria<br>Therefo<br>excepti<br>Sectior<br>study,<br>questic<br>Group's | does not allow for the issuance of waivers to any protocol specified ( <a href="http://ctep.cancer.gov/protocolDevelopment/policies_deviations.htm">http://ctep.cancer.gov/protocolDevelopment/policies_deviations.htm</a> ). Ore, all eligibility criteria listed in Section 2 must be met, without ion. The registration of individuals who do not meet all criteria listed in a 2 can result in the participant being censored from the analysis of the and the citation of a major protocol violation during an audit. All ons regarding clarification of eligibility criteria must be directed to the sexecutive Officer ( <a href="EA.Execofficer@jimmy.harvard.edu">EA.Execofficer@jimmy.harvard.edu</a> ) or the sexegulatory Officer ( <a href="EA.Execofficer@jimmy.harvard.edu">EA.Execofficer@jimmy.harvard.edu</a> ). |
| | NOTE: | l | been re | ions may use the eligibility checklist as source documentation if it has eviewed, signed, and dated prior to registration/randomization by the physician. |
| | NOTE: | , | All pati | ents must have signed the relevant treatment consent form. |
| Rev. 8/15 | 2.1 | Eligi | ibility C | <u>Criteria</u> |
| Rev. Add13 | | 2.1. | 1 | Patients must be positive for translocation or inversion events involving the ROS1 gene via the MATCH Master Protocol and described in Appendix IV. See <u>Appendix IV</u> for information on the ROS1 translocations and inversions and corresponding LOEs. |
| Rev. 2/16 | | 2.1. | 2 | Patients must not have NSCLC with ROS1 rearrangements. |
| Rev. 8/15 | | 2.1. | 3 | Patients with a history of interstitial lung disease or pneumonitis are excluded. |
| Rev. 2/16 | | 2.1.4 | 4 | Patient must fulfill all eligibility criteria outlined in Section 3.1 of the MATCH Master Protocol (excluding Section 3.1.6) at the time of registration to treatment step (Step 1, 3, 5, 7). |
| Rev. 8/15 | | 2.1. | 5 | Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block). |
| | | | | Date of ECG: |
| | | 2.1.0 | 6 | Patients must not have known hypersensitivity to crizotinib or compounds of similar chemical or biologic composition. |

| EAY131-G | j |
|----------------------------------|---|
| Version Date: January 25, 2019 | • |
| MCI Undate Date: August 12, 2018 | = |

| <br>2.1.7 | Patients using drugs or foods that are known poinhibitors or inducers will be excluded (See App | |
|---|---|---|
| 2.1.8 | Patients must not have had prior therapy with a including crizotinib, ceritinib, foretinib, cabozant ASP3026, WZ-5-126, TAE684, KIST301072, KIPF-06463922, RXDX-101 and PF-3922 | inib, AP26113, |
| | Physician Signature | Date |

This signature line is provided for use by institutions wishing to use the eligibility checklist as source documentation. **OPTIONAL:** 

NCI Update Date: August 12, 2015

#### 3. Criztonib Treatment Plan

#### 3.1 <u>Administration Schedule</u>

Study Drug: Crizotinib

Crizotinib capsules, 250 mg, will be administered orally twice daily on a continuous daily dosing schedule, ie, no break in dosing. Crizotinib should be taken approximately 12 hours apart and without regard to meals. Cycles are defined in 28-day periods to facilitate scheduling of visits and assessments.

Patients should be instructed that if they vomit after taking a dose, then they must not "make it up" with an extra dose, but instead, resume subsequent doses as prescribed. Any missed dose may be taken up to 6 hours prior to the next scheduled dose, otherwise it should be skipped and dosing resumed with subsequent doses.

#### 3.2 Adverse Event Reporting Requirements

The Adverse Event Reporting Requirements for all EAY131 subprotocols are outlined in the MATCH MASTER protocol. Please refer to those guidelines when determining if an event qualifies as a Serious Adverse Event (SAE) and requires expedited reporting via CTEP's Adverse Event Reporting System (CTEP-AERS).

In addition, the following section outlines agent specific requirements and must be followed to ensure all reporting requirements are met.

3.2.1 Additional adverse event reporting instructions, requirements and instructions for protocol EAY131 – Subprotocol G

#### **Additional Instructions**

For instructions on how to specifically report events that result in persistent or significant disability/incapacity, congenital anomaly, or birth defect events via CTEP-AERS, please contact the AEMD Help Desk at <a href="mailto:aemd@tech-res.com">aemd@tech-res.com</a> or 301-897-7497. This will need to be discussed on a case-by-case basis.

### **EAY131-** Subprotocol G specific expedited reporting requirements:

• Pregnancies: Pregnancies and suspected pregnancies (including a positive or inconclusive pregnancy test, regardless of age or disease state) occurring while the subject is on Crizotinib, or within 28 days of the subject's last dose of Crizotinib, are considered immediately reportable events. The pregnancy, suspected pregnancy, or positive/ inconclusive pregnancy test must be reported via CTEP-AERS within 24 hours of the Investigator's knowledge. Please refer to Appendix VIII in MATCH Master protocol for detailed instructions on how to report the occurrence of a pregnancy as well as the outcome of all pregnancies.

### EAY131 – Subprotocol G specific expedited reporting exceptions:

For subprotocol G, the adverse events listed below **do not** require expedited reporting via CTEP-AERS:

If an AE meets the reporting requirements of the protocol, and it
is listed on the SPEER, it should <u>ONLY</u> be reported via CTEPAERS if the grade being reported exceeds the grade listed in
the parentheses next to the event.

#### 3.2.2 Second Primary Cancer Reporting Requirements

All cases of second primary cancers, including acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS), that occur following treatment on NCI-sponsored trials must be reported to ECOG-ACRIN using Medidata Rave

- A <u>second malignancy</u> is a cancer that is UNRELATED to any prior anti-cancer treatment (including the treatment on this protocol). Second malignancies require ONLY routine reporting as follows:
  - Complete a Second Primary Form in Medidata Rave within 14 days.
  - 2. Upload a copy of the pathology report to ECOG-ACRIN via Medidata Rave confirming the diagnosis.
  - If the patient has been diagnosed with AML/MDS, upload a copy of the cytogenetics report (if available) to ECOG-ACRIN via Medidata Rave.
- A <u>secondary malignancy</u> is a cancer CAUSED BY any prior anticancer treatment (including the treatment on this protocol).
   Secondary malignancies require both routine and expedited reporting as follows:
  - Complete a Second Primary Form in Medidata Rave within 14 days
  - 2. Report the diagnosis via CTEP-AERS at <a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>
    Report under a.) leukemia secondary to oncology
    chemotherapy, b.) myelodysplastic syndrome, or c.)
    treatment related secondary malignancy
  - 3. Upload a copy of the pathology report to ECOG-ACRIN via Medidata Rave and submit a copy to NCI/CTEP confirming the diagnosis.
  - If the patient has been diagnosed with AML/MDS, upload a copy of the cytogenetics report (if available) to ECOG-ACRIN via Medidata Rave and submit a copy to NCI/CTEP.

**NOTE:** The Second Primary Form and the CTEP-AERS report should not be used to report recurrence or development of metastatic disease.

**NOTE:** If a patient has been enrolled in more than one NCI-

sponsored study, the Second Primary Form must be submitted for the most recent trial. ECOG-ACRIN must be provided with a copy of the form and the associated pathology report and cytogenetics report (if available) even if ECOG-ACRIN was not the patient's most recent trial.

**NOTE:** Once data regarding survival and remission status are no

longer required by the protocol, no follow-up data should be submitted via CTEP-AERS or by the Second Primary

Form.

Rev. 5/16 Rev. 8/17 Rev. Add18

#### 3.3 Comprehensive Adverse Events and Potential Risks List (CAEPR) for Crizotinib (PF-02341066, NSC 749005)

The Comprehensive Adverse Events and Potential Risks list (CAEPR) provides a single list of reported and/or potential adverse events (AE) associated with an agent using a uniform presentation of events by body system. In addition to the comprehensive list, a subset, the Specific Protocol Exceptions to Expedited Reporting (SPEER), appears in a separate column and is identified with bold and italicized text. This subset of AEs (SPEER) is a list of events that are protocol specific exceptions to expedited reporting to NCI (except as noted below). Refer to the 'CTEP, NCI Guidelines: Adverse Event Reporting Requirements' http://ctep.cancer.gov/protocolDevelopment/electronic applications/docs/aequide lines.pdf for further clarification. Frequency is provided based on 2058 patients. Below is the CAEPR for Crizotinib (PF-02341066).

NOTE:

If an AE meets the reporting requirements of the protocol, and it is listed on the SPEER, it should **ONLY** be reported via CTEP-AERS if the grade being reported exceeds the grade listed in the parentheses next to the event in the SPEER.

Version 2.3, October 30, 2018<sup>1</sup>

| Relati | Specific Protocol<br>Exceptions to<br>Expedited Reporting<br>(SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| BLOOD AND LYMPHAT | C SYSTEM DISORDERS | | |
| | Anemia | | Anemia (Gr 2) |
| | | Febrile neutropenia | |
| CARDIAC DISORDERS | | | |
| | | Heart failure | |
| | Sinus bradycardia | | |
| ENDOCRINE DISORDER | RS | | |
| | | Testosterone deficiency | |
| EYE DISORDERS | | | |
| Eye disorders - Other (vision disorders) <sup>2</sup> | | | Eye disorders - Other<br>(vision disorders) <sup>2</sup><br>(Gr 2) |
| Periorbital edema | | | Periorbital edema (Gr 2) |
| GASTROINTESTINAL D | ISORDERS | | |
| | Abdominal pain | | Abdominal pain (Gr 2) |
| | | Colonic perforation | |
| Constipation | | | Constipation (Gr 2) |
| Diarrhea | | | Diarrhea (Gr 2) |
| | Dyspepsia | | |
| | | Esophageal ulcer | |
| | | Esophagitis | |

| A(<br>Relatio | Specific Protocol<br>Exceptions to<br>Expedited Reporting<br>(SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| | Mucositis oral | | |
| Nausea | | | Nausea (Gr 2) |
| Vomiting | | | Vomiting (Gr 2) |
| GENERAL DISORDERS A | AND ADMINISTRATION SI | TE CONDITIONS | |
| Edema face | | | Edema face (Gr 2) |
| Edema limbs | | | Edema limbs (Gr 2) |
| Fatigue | | | Fatigue (Gr 2) |
| Generalized edema | | | Generalized edema<br>(Gr 2) |
| Localized edema | | | Localized edema (Gr 2) |
| HEPATOBILIARY DISORI | DERS | | |
| | | Hepatic failure | |
| | | Hepatobiliary disorders - Other (hepatotoxicity) | |
| INFECTIONS AND INFES | | | |
| | Upper respiratory infection | | |
| INVESTIGATIONS | 1 | | |
| | Alanine aminotransferase increased | | Alanine<br>aminotransferase<br>increased (Gr 2) |
| | Alkaline phosphatase increased | | |
| | Aspartate aminotransferase increased | | Aspartate<br>aminotransferase<br>increased (Gr 2) |
| | | Blood bilirubin increased | |
| | Creatinine increased | | |
| | | Electrocardiogram QT corrected interval prolonged | |
| | Lymphocyte count decreased | | |
| Neutrophil count decreased | | | Neutrophil count<br>decreased (Gr 2) |
| | White blood cell decreased | | White blood cell<br>decreased (Gr 2) |
| METABOLISM AND NUT | RITION DISORDERS | | |
| | Anorexia | | Anorexia (Gr 2) |
| MUSCULOSKELETAL AN | ID CONNECTIVE TISSUE I | DISORDERS | |
| | Muscle cramp | | |

| Ad<br>Relatio | Specific Protocol<br>Exceptions to<br>Expedited Reporting<br>(SPEER) | | |
|---|---|---|---|
| Likely (>20%) | Less Likely (<=20%) | Rare but Serious (<3%) | |
| NERVOUS SYSTEM DISC | ORDERS | | |
| | Dizziness | | Dizziness (Gr 2) |
| | Dysgeusia | | Dysgeusia (Gr 2) |
| | Nervous system disorders - Other (neuropathy) <sup>3</sup> | | Nervous system<br>disorders - Other<br>(neuropathy)³ (Gr 2) |
| | | Syncope | |
| RENAL AND URINARY D | SORDERS | | |
| | | Renal and urinary<br>disorders - Other (renal<br>cyst) | |
| RESPIRATORY, THORAC | | | |
| | | Pneumonitis | |
| SKIN AND SUBCUTANEO | SKIN AND SUBCUTANEOUS TISSUE DISORDERS | | |
| | Rash <sup>4</sup> | | |

<sup>&</sup>lt;sup>1</sup>This table will be updated as the toxicity profile of the agent is revised. Updates will be distributed to all Principal Investigators at the time of revision. The current version can be obtained by contacting <a href="PIO@CTEP.NCI.NIH.GOV">PIO@CTEP.NCI.NIH.GOV</a>. Your name, the name of the investigator, the protocol and the agent should be included in the e-mail.

<sup>&</sup>lt;sup>2</sup>Vision disorders may include the following: Chromatopsia, Diplopia, Halo vision, Photophobia, Photopsia, Vision blurred, Visual acuity reduced, Visual brightness, Visual impairment, Vitreous floaters, and Visual perseveration.

<sup>&</sup>lt;sup>3</sup>Neuropathy may include the following: Acute polyneuropathy, Amyotrophy, Areflexia, Autoimmune neuropathy, Autonomic failure syndrome, Autonomic neuropathy, Axonal neuropathy, Biopsy peripheral nerve abnormal, Burning feet syndrome, Burning sensation, Decreased vibratory sense, Demyelinating polyneuropathy, Dysesthesia, Electromyogram abnormal, Formication, Gait disturbance, Genital hypoesthesia, Guillain-Barre syndrome, Hyperesthesia, Hypoesthesia, Hyporeflexia, Hypotonia, Ischemic neuropathy, Loss of proprioception, Miller Fisher syndrome, Mononeuritis, Mononeuropathy, Mononeuropathy multiplex, Motor dysfunction, Multifocal motor neuropathy, Muscle atrophy, Muscular weakness, Myelopathy, Nerve conduction studies abnormal, Nerve degeneration, Neuralgia, Neuritis, Neuromuscular toxicity, Neuromyopathy, Neuropathy peripheral, Neuropathy vitamin B6 deficiency, Neurotoxicity, Paresthesia, Peripheral motor neuropathy, Peripheral nerve lesion, Peripheral nerve palsy, Peripheral nervous system function test abnormal, Peripheral sensorimotor neuropathy, Peripheral sensory neuropathy, Peroneal muscular atrophy, Peroneal nerve palsy, Phrenic nerve paralysis, Polyneuropathy, Polyneuropathy chronic, Polyneuropathy idiopathic progressive, Radiation neuropathy, Sensorimotor disorder, Sensory disturbance, Sensory loss, Skin burning sensation, Temperature perception test decreased, Tinel's sign, Toxic neuropathy, and Ulnar neuritis.

<sup>&</sup>lt;sup>4</sup>Treatment-related rash may include erythematous rash, rash maculo-papular, and pruritus.

Adverse events reported on crizotinib (PF-02341066) trials, but for which there is insufficient evidence to suggest that there was a reasonable possibility that crizotinib (PF-02341066) caused the adverse event:

**BLOOD AND LYMPHATIC SYSTEM DISORDERS** - Blood and lymphatic system disorders - Other (basophilia); Disseminated intravascular coagulation; Eosinophilia; Leukocytosis

**CARDIAC DISORDERS** - Atrial fibrillation; Cardiac arrest; Chest pain - cardiac; Myocarditis; Pericardial effusion; Supraventricular tachycardia

EYE DISORDERS - Cataract; Optic nerve disorder; Papilledema

**GASTROINTESTINAL DISORDERS** - Colitis; Dysphagia; Gastric ulcer; Gastroesophageal reflux disease; Gastrointestinal disorders - Other (gastrointestinal amyloidosis); Ileus

**GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS** - Fever; General disorders and administration site conditions - Other (failure to thrive); Malaise; Non-cardiac chest pain

**HEPATOBILIARY DISORDERS** - Hepatobiliary disorders - Other (cholestasis); Hepatobiliary disorders - Other (hepatitis)

**IMMUNE SYSTEM DISORDERS** - Autoimmune disorder

**INFECTIONS AND INFESTATIONS** - Abdominal infection; Infections and infestations - Other (peridiverticular abscess); Kidney infection; Lung infection; Sepsis; Skin infection; Urinary tract infection

**INJURY, POISONING AND PROCEDURAL COMPLICATIONS** - Injury, poisoning and procedural complications - Other (traumatic lung injury); Spinal fracture; Wound complication

**INVESTIGATIONS** - Blood lactate dehydrogenase increased; CPK increased; GGT increased; Investigations - Other (monocyte count increased); Investigations - Other (platelet count increased); Platelet count decreased

**METABOLISM AND NUTRITION DISORDERS** - Dehydration; Hyperglycemia; Hyperkalemia; Hypermagnesemia; Hypertriglyceridemia; Hypoalbuminemia; Hypocalcemia; Hypokalemia; Hyponatremia; Hypophosphatemia; Metabolism and nutrition disorders - Other (hypoproteinemia)

MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS - Arthralgia;

Musculoskeletal and connective tissue disorder - Other (myopathy); Myalgia; Pain in extremity

**NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)** - Treatment related secondary malignancy: Tumor hemorrhage

**NERVOUS SYSTEM DISORDERS** - Intracranial hemorrhage; Ischemia cerebrovascular; Pyramidal tract syndrome; Seizure; Stroke

PREGNANCY, PUERPERIUM AND PERINATAL CONDITIONS - Pregnancy loss

PSYCHIATRIC DISORDERS - Confusion; Delirium; Euphoria

**RENAL AND URINARY DISORDERS** - Acute kidney injury; Hematuria; Renal calculi; Urinary retention

**RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS** - Bronchopulmonary hemorrhage; Dyspnea; Pleural effusion; Respiratory failure; Respiratory, thoracic and mediastinal disorders - Other (pneumomediastinum); Respiratory, thoracic and mediastinal disorders - Other (respiratory distress)

**SKIN AND SUBCUTANEOUS TISSUE DISORDERS** - Skin and subcutaneous tissue disorders - Other (drug eruption)

EAY131-G

Version Date: January 25, 2019 NCI Update Date: August 12, 2015

**VASCULAR DISORDERS** - Hematoma; Hypotension; Phlebitis; Thromboembolic event; Vasculitis

**NOTE:** Crizotinib (PF-02341066) in combination with other agents could cause an

exacerbation of any adverse event currently known to be caused by the other agent, or the combination may result in events never previously associated with either

agent.

EAY131-G

Version Date: January 25, 2019 NCI Update Date: August 12, 2015

#### 3.4 Dose Modifications

All toxicity grades below are described using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP website (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>).

Patients will be monitored closely for toxicity and the dose of crizotinib may be adjusted as indicated in Table 3.5. Intrapatient dose reduction by 1, and if needed, 2 dose level(s) will be allowed depending on the type and severity of toxicity encountered.

| Dose Level | Crizotinib Dose |
|------------|-----------------|
| 1 | 250mg BID |
| -1 | 200mg BID |
| -2 | 250mg Daily |

Patients requiring more than 2 dose reductions due to treatment-toxicity will be removed from treatment. Patients requiring treatment to be held for >4 weeks will be taken off treatment.

Table 3.5 Crizotinib Dose Modifications for Treatment-Related Toxicity

| Toxicity | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
|---|---|---|---|---|
| Non- hematologic General (except<br>as noted below), eg, neuropathy,<br>edema (including peripheral<br>edema and localized edema),<br>fatigue, and skin rash (including<br>erythematous, macular, papular,<br>and pruritic rash) | Continue at the same dose level. | Continue at the same dose level. | Withhold dose until toxicity is Grade ≤ 1, or has returned to baseline, then resume treatment at the same dose level or reduce the dose by 1 level at the discretion of the investigator.* | Withhold dose until toxicity is Grade ≤ 1, or has returned to baseline, then reduce the dose by 1 level and resume treatment, or discontinue at the discretion of the investigator*. |
| ALT elevation with total bilirubin < 2 X ULN (in the absence of cholestasis or hemolysis) § | Continue at the same dose level. | Continue at the same dose level. Obtain repeat ALT and total bilirubin when symptomatic or within 7 days. | Withhold dose until toxicity is grade 1, or has returned to baseline, then resume treatment by reducing the dose by one dose level. If Grade 3 ALT elevation recurs reduce further (at most by 2 dose levels from initial dose level). If recurrence at dose level -2, discontinue permanently. If Grade 3 ALT elevation does not recur after at least 4 weeks, the dose may be escalated by single dose level increments up to the initial dose level. | See Grade 3. |
| ALT elevation concurrent with total bilirubin elevation ≥ 2 X ULN (in the absence of cholestasis or hemolysis) | Continue at the same dose level. Obtain repeat ALT and total bilirubin within 48 hours. | Discontinue<br>treatment and<br>do not retreat | Discontinue treatment and do not retreat | Discontinue treatment and do not retreat |
| Left ventricular systolic dysfunction | Continue at the same dose level | Continue at the same dose level | Discontinue treatment and do not retreat | Discontinue treatment and do not retreat |

| Prolonged QTc | Continue at the same dose level | Assess electrolytes and concomitant medications. Correct any electrolyte or magnesium abnormalities | Interrupt crizotinib until recovery to baseline. Assess and correct electrolytes and concomitant medications. Resume treatment by reducing the dose by one dose level, unless an alternative cause for QTc prolongation is found and corrected, resume at the same dose level. | Discontinue treatment and do not retreat |
|---|---|---|---|---|
| Pneumonitis (in absence of disease progression, pulmonary embolism, positive cultures or radiation effect) | Discontinue treatment and do not retreat | Discontinue<br>treatment and<br>do not retreat | Discontinue treatment and do not retreat | Discontinue treatment and do not retreat |
| Visual disturbance | Continue at the same dose level. Repeat ophthalmologic examination+ | Continue at the same dose level. Repeat ophthalmologic examination+ | Interrupt crizotinib until recovery. Repeat ophthalmologic examination+. Resume treatment by reducing by one dose level. | Discontinue treatment and do not retreat. Repeat ophthalmologic examination+. |
| Hematologic (excluding lymphopenia**) | Continue at the same dose level. | Continue at the same dose level. | Withhold dose until toxicity is Grade ≤ 2, or has returned to baseline, then resume treatment at the same dose level or reduce by 1 level after discussion with the study chair**/***. | Withhold dose until toxicity is Grade ≤ 2, or has returned to baseline, then reduce the dose by 1 level and resume treatment**. |
| Hypophosphatemia or hyperuricemia* | Continue at the same dose level | Continue at the same dose level | Continue at the same dose level at investigator discretion | Discontinue treatment until resolution to grade 3 or lower |

<sup>\*</sup> Patients who develop Grade 3 hyperuricemia or Grade 3 hypophosphatemia without clinical symptoms may continue study treatment without interruption at the discretion of the investigator. Nausea, vomiting or diarrhea must persist at Grade 3 or 4 despite maximal medical therapy, to require dose modification.

+ Ophthalmologic examination includes visual acuity and slit lamp and should be performed by an ophthalmologist.

<sup>\*\*</sup> Patients who develop Grade 3 or 4 lymphopenia without other dose-limiting events (eg, opportunistic infection) may continue study treatment without interruption.

<sup>\*\*\*</sup> Patients entering with platelet counts > 30,000 (to < 50,000/µL) will be monitored for drug related decreases at which point dose modifications will be discussed with the Sponsor

<sup>§</sup> Patients entering with ALT and/or AST ≥5 x ULN (ie, Grade ≥3) due to underlying malignancy will be monitored for potential drug related increases at which point dose modifications will be discussed with the Sponsor (Note: this option does not apply for France).

#### 3.5 Supportive Care

All supportive measures consistent with optimal patient care will be given throughout the study.

- 3.5.1 Nausea and emesis: For nausea and vomiting, treat with standard anti-emetics such as prochloroperazine or ondansetron. Patients should be counseled that taking the medication with food may reduce nausea. The use of prophylactic antiemetics should be considered. Given the potential for ondansetron to increase QTc prolongation. review baseline QTc EKG prior to initiation of ondansetron and consider follow up EKGs on treatment.
- 3.5.2 Diarrhea: For grade 1 diarrhea, symptomatic care such as loperamide (Imodium) or no intervention at investigator judgment. For grade 2 diarrhea, loperamide (4 mg at first onset, then 2 mg every 2-4 hrs until symptom free for 12 hours). See Section 3.4 for instructions on dose modifications.

3.5.3 Bradycardia:

Rev. 8/15

| Bradycardia<br>(heart rate less<br>than 60 beats<br>per minute) | Continue at the same dose level. | to heart rate ≥ 60. | Same as for<br>Grade 2<br>bradycardia. | Permanently discontinue if no contributing concomitant medication is identified. |
|---|---|---|---|---|
| | | anti-hypertensive medications. If contributing concomitant medication is identified and discontinued, or its dose is adjusted, resume at previous dose upon recovery to Grade ≤ 1 or to heart rate ≥ 60. If no contributing concomitant medication is identified, or if contributing concomitant medications are not discontinued or dose modified, resume at reduced dose upon recovery to Grade ≤ 1 or to heart rate ≥60. | | If contributing concomitant medication is identified and discontinued, or its dose is adjusted, resume at 250 mg once daily upon recovery to Grade ≤ 1 or to heart rate ≥ 60, with frequent monitoring. Permanently discontinue for recurrence. |

- 3.5.4 Pneumonitis/pneumonia: Investigators must evaluate thoroughly patients who demonstrate potential signs or symptoms of pneumonitis or pneumonia. If a patient has a potential diagnosis of pneumonitis or drug-related lung injury, the following evaluations/procedures should be considered to assist or exclude the diagnosis of pneumonitis:
  - Evaluate for pneumonia: Pneumonia would be supported by clinical symptoms/signs of infection, including fever, leukocytosis, productive cough, characteristic radiologic findings, and most importantly, documentation of microbiology studies (sputum gram/stain and culture, blood cultures). Pneumonia should be treated with the appropriate antibiotics and supportive care. Many of these symptoms/signs may be seen in pneumonitis, but in this case, all microbiological studies would be negative (including possibly bronchoscopy for specimens).

- Sputum gram stain and culture (induced sputum if needed), to evaluate for bacterial, viral, fungal, protozoal, and mycobacterial infections
- Blood cultures if febrile
- Thoracentesis if pleural fluid is present (examined for the same pathogens as in 3.6.4.1)
- Bronchoscopy with bronchoalveolar lavage (BAL) if appropriate.
   BAL fluid should be sent for culture and cytology (same pathogens as 3.6.4.1)
- Lung biopsy if appropriate and necessary to distinguish between pneumonia and pneumonitis
- BNP levels to evaluate for heart failure
- If clinically appropriate, particularly if pneumonia can be ruled out, high dose corticosteroid treatment should be initiated. Should the event be fatal, an autopsy is recommended to confirm/exclude the diagnosis.
- 3.5.5 Renal cysts: Complex renal cysts have been reported in some patients treated with crizotinib. These cysts may be symptomatic or asymptomatic, and typically develop between 2 and 6 months after starting crizotinib. The precise nature and significance of these cysts is unclear. However, complex renal cysts can be associated with renal malignancy, so consultation with a urologist is recommended. Urinalysis should be performed if renal cysts are detected, and followed on Day 1 of each cycle thereafter. Urine reflex microscopy is required if the urinalysis demonstrates blood or protein.
- 3.5.6 Hypogonadism: For males reporting symptoms of hypogonadism (fatigue, sexual dysfunction, decreased libido, mood or sleep disorder, gynecomastia), a panel of blood tests should be drawn, including total testosterone, free testosterone, and sex-hormone binding globulin (SHBG). If free testosterone is low, consultation with endocrinology is recommended for possible testosterone supplementation

#### 3.6 Duration of Agent-specific treatment

In the absence of treatment delays due to adverse event(s), treatment may continue until one of the following criteria applies:

- Extraordinary Medical Circumstances: If at any time the constraints of this
  protocol are detrimental to the patient's health, protocol treatment should be
  discontinued. In this event submit forms according to the instructions in the
  MATCH Forms Packet.
- Patient withdraws consent.
- Patient experiences unacceptable toxicity.
- Non-protocol therapies are administered.
- Disease progression

#### 3.7 Duration of Follow-Up

Refer to the MATCH Master Protocol for specifics on the duration of follow-up.

#### Rev. 12/16 **4. Study Parameters**

Rev. 8/15, 2/16 Rev. 3/17

#### 4.1 <u>Therapeutic Parameters for Crizotinib Treatment</u>

**NOTE:** In addition to the study parameters listed in the MATCH Master Protocol at Step 0, the below parameters

must also be performed for patients on Crizotinib treatment.

**NOTE:** All assessments required prior to registration to treatment should be done ≤ 4 weeks prior to registration to

Steps 1, 3, 5, 7, excluding the radiologic evaluation and electrocardiogram (ECG).

Rev. 2/16

| T1/A | Prior to Pogistration | Treatn | nent | End of | |
|---|---|---|---|---|---|
| Test/Assessment | Prior to Registration to Treatment | Every Cycle, prior to treatment | Every 2 Cycles | Treatment | Follow Up <sup>F</sup> |
| H&P, Weight, Vital signs <sup>A</sup> | X | X <sub>1</sub> | | | Х |
| Performance status | X | X <sub>1</sub> | | | Х |
| CBC w/diff, plts <sup>B</sup> | X | X <sub>1</sub> | | | Х |
| Serum chemistry <sup>B</sup> | X | X <sub>1</sub> | | | Х |
| Radiologic evaluation <sup>D</sup> | X | | XD | | X <sup>F</sup> |
| β-HCG <sup>c</sup> | X | | | | |
| Toxicity Assessment <sup>G</sup> | | X | | Х | X <sup>F</sup> |
| Pill Count/Diary <sup>H</sup> | | X | | Х | |
| ECG <sup>K</sup> | X | Χι | | | |
| Tumor biopsy and blood sample for MATCH<br>Master protocol <sup>E</sup> | | | Х | Х | |

A. History and physical, including vital signs and weight at the start of each cycle (up to 3 days before start of new cycle).

Rev. 2/16 Rev. 5/16

- B. Albumin, alkaline phosphatase, total bilirubin, bicarbonate, BUN, calcium, creatinine, glucose, phosphorus, potassium, SGOT[AST], SGPT[ALT], sodium, magnesium and serum tumor markers (including LDH, PSA if appropriate). For eligibility purposes, participants with creatinine levels above institutional normal, Cockcroft-Gault will be used to calculate creatinine clearance. CBC w/diff, platelets and serum chemistries should be performed on cycle 1, day 1 (or up to 7 days prior), and at the start of each subsequent cycle (up to 3 days before start of new cycle). CBC with differential will be performed more frequently in patients with grade 4 neutropenia or thrombocytopenia until resolution to ≤ grade 3. CBC and serum chemistries are only required in follow-up until values return to pre-treatment levels or until progressive disease.
- <sup>C.</sup> Blood pregnancy test (women of childbearing potential) required prior to beginning treatment.

Rev. 2/16

Disease measurements are repeated every 2 cycles for first 26 cycles, and every 3 cycles thereafter until PD or start of another MATCH treatment step. The baseline evaluation should be performed as closely as possible to the beginning of treatment and never more than 6 weeks before registration to treatment step. For multiple myeloma patients, please refer to Section 6.4 of the MATCH Master Protocol for additional information

on myeloma response criteria and the required disease assessments. Documentation (radiologic) must be provided for patients removed from study for progressive disease.

- Rev. Add13 E. Additional blood specimens and/or biopsies are to be submitted from consenting patients per Section 9.3.2 of the MATCH Master Protocol. Submit at the following time points, as applicable:
  - Blood specimens are to be submitted at the end of Cycle 2 (prior to start of Cycle 3 treatment). If patient progresses or treatment is discontinued prior to Cycle 3, collect the blood at that time instead. On-treatment kits for blood sample collections will be automatically shipped to sites upon registration to the treatment step.
  - Screening biopsies for additional aMOI assessments after registration to appropriate screening step, if applicable (Step 2 or Step 4).

Rev. 2/16

At end of all MATCH study treatments, blood specimens and/or research biopsy after consent and registration to Step 8

Please refer to Section 4 of the MATCH Master Protocol to determine whether the patient proceeds to the next screening step or to follow-up (with a potential end of treatment biopsy for research purposes on Step 8). Samples are to be submitted as outlined in Section 9 of the MATCH Master Protocol, To order Step 2/4 Screening or Step 8 kits, complete the EAY131 Collection and Shipping Kit Order Form (See Appendix XII of the MATCH Master Protocol) and fax to 713-563-6506.

- F. Every 3 months if patient is < 2 years from study entry, and every 6 months for year 3. Toxicity assessments and radiologic evaluations are not required to be done during Follow Up if progression has been previously reported; however if an adverse event occurs post treatment that meets the SAE reporting requirements, it still must be reported via CTEP-AERS, even if progression has occurred.
- G. Site personnel should evaluate for toxicity and discuss treatment compliance with the patient in order to ensure the medication is taken correctly; this evaluation may be conducted by telephone or in person. The Toxicity Assessment is not required prior to Cycle 1, but is required every subsequent cycle.
- H. The pill calendar will be collected at the end of every cycle. The Pill Count/Diary is not required prior to Cycle 1, but is required every subsequent cycle.
- 1. As clinically indicated.
- J. For Cycle 1, if the following tests/assessments occurred within 7 days of Day 1, they do not need to be repeated at this timepoint: H&P, Weight, Vital Signs: Performance Status: CBC w/diff, plts; Serum chemistry: Concomitant Medications.
- K. Within 8 weeks of treatment assignment.

#### Rev. Add13 5. Drug Formulation and Procurement

This information has been prepared by the ECOG-ACRIN Pharmacy and Nursing Committees.

#### **Availability**

Rev. 8/15

NO STARTER SUPPLIES MAY BE ORDERED. Subjects must be enrolled and assigned to the treatment subprotocol prior to submitting the clinical drug request to PMB.

Drug Ordering: NCI supplied agents may be requested by eligible participating Investigators (or their authorized designee) at each participating institution. Pharmaceutical Management Branch (PMB) policy requires that drug be shipped directly to the institution where the patient is to be treated. PMB does not permit the transfer of agents between institutions (unless prior approval from PMB is obtained – see general information) The CTEP-assigned protocol number must be used for ordering all CTEP-supplied investigational agents. The eligible participating investigators at each participating institution must be registered with CTEP, DCTD through an annual submission of FDA Form 1572 (Statement of Investigator), NCI Biosketch, Agent Shipment Form, and Financial Disclosure Form (FDF). If there are several participating investigators at one institution, CTEP-supplied investigational agents for the study should be ordered under the name of one lead investigator at that institution.

Submit agent requests through the PMB Online Agent Order Processing (OAOP) application (<a href="https://ctepcore.nci.nih.gov/OAOP">https://ctepcore.nci.nih.gov/OAOP</a>). Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account (<a href="https://ctepcore.nci.nih.gov/iam/">https://ctepcore.nci.nih.gov/iam/</a>) and the maintenance of an "active" account status, a "current" password, and an active person registration status.

#### NCI Supplied Agent(s) – General Information

Questions about drug orders, transfers, returns, or accountability should be addressed to the PMB by calling 240-276-6575 Monday through Friday between 8:30 AM and 4:30 PM Eastern Time or email <a href="mailto:PMBAfterHours@mail.nih.gov">PMBAfterHours@mail.nih.gov</a> anytime.

**Drug Returns:** All undispensed drug supplies should be returned to the PMB. When it is necessary to return study drug (e.g., sealed bottles remaining when PMB sends a stock recovery letter), investigators should return the study drug to the PMB using the NCI Return Agent Form available on the NCI home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>).

**Drug Accountability:** The investigator, or a responsible party designated by the investigator, must maintain a careful record of the receipt, disposition, and return of agent received from the PMB using the NCI Investigational Agent Accountability Record Form for Oral Agents available on the NCI home page (<a href="http://ctep.cancer.gov">http://ctep.cancer.gov</a>). Maintain separate NCI Investigational Agent Accountability Records for each agent, strength, formulation and ordering investigator.

Rev. 12/16

Rev. 3/17

Investigator Brochure Availability: The current versions of the IBs for PMB-supplied agents will be accessible to site investigators and research staff through the PMB Online Agent Order Processing (OAOP) application. Access to OAOP requires the establishment of a CTEP Identity and Access Management (IAM) account and the maintenance of an "active" account status, a "current" password, and active person

registration status. Questions about IB access may be directed to the PMB IB coordinator at IBCoordinator@mail.nih.gov.

#### 5.1 <u>Crizotinib (NSC #749005)</u>

#### 5.1.1 Other Names

Xalkori®, PF-02341066

#### 5.1.2 Classification

**ALK** inhibitor

#### 5.1.3 Mode of Action

Crizotinib is a selective ATP-competitive small –molecule inhibitor of anaplastic lymphoma kinase (ALK), c-Met/hepatocyte growth factor receptor (HGFR) and Recepteur d'Origine Nantais (RON), and ROS1 receptor tyrosine kinases and their oncogenic variants. Translocations of these genes can result in expression of oncogenic fusion proteins that contribute to increased cell proliferation and survival. Antitumor efficacy of crizotinib is correlated to pharmacodynamic inhibition of phosphorylation of ALK fusion variants or c-Met/HGFR in tumors in vivo.

#### 5.1.4 Storage and Stability

**Storage:** Store at room temperature 20° to 25° C (68° to 77° F).

**Stability:** Shelf life is consistent with commercially-labeled product.

#### 5.1.5 Dose Specifics

Crizotinib capsules, 250 mg, will be administered orally twice daily on a continuous daily dosing schedule.

#### 5.1.6 Preparation

Pfizer supplies and PMB, CTEP, DCTD distributes commercially-labeled crizotinib as 200 mg (size 1, white opaque body and pink opaque cap, with "Pfizer" on the cap and "CRZ 200" on the body) and 250 mg (size 0, pink opaque body and cap, with "Pfizer" on the cap and "CRZ 250 on the body) hard gelatin capsules. Each bottle contains 60 capsules.

Excipients include colloidal silicon dioxide, microcrystalline cellulose, anhydrous dibasic calcium phosphate, sodium starch glycolate, magnesium stearate, and hard gelatin capsule shells as inactive ingredients.

The pink opaque capsule shell components contain gelatin, titanium dioxide, and red iron oxide. The white opaque capsule shell components contain gelatin, and titanium dioxide. The printing ink contains shellac, propylene glycol, strong ammonia solution, potassium hydroxide, and black iron oxide.

#### 5.1.7 Route of Administration

Oral. Take with or without food.

Rev. 12/16 Rev.Add13

#### 5.1.8 Incompatibilities

Crizotinib is primarily metabolized by CYP 3A4/5 with minor contributions from CYP2C8, CYP2C19, and CYP2D6. Avoid concomitant use of strong CYP3A inhibitors and inducers. Use of potent CYP3A inducers should be avoided for at least 12 days prior to the first dose of crizotinib. Use of strong CYP3A inhibitors should be avoided for at least 7 days prior to the first dose of crizotinib. Exercise caution with concomitant use of moderate CYP3A inhibitors. Crizotinib moderately inhibits CYP3A4 in a time-dependent fashion. Use caution with patients who receive CYP3A4 substrates with a narrow therapeutic index.

Crizotinib is an inhibitor of CYP2B6 in vitro. Use caution with coadministered drugs that are predominantly metabolized by CYP2B6.

Studies demonstrate that crizotinib is a substrate of P-gp and a weak BCRP inhibitor, however the potential to cause drug-drug interactions at therapeutic doses is low. Crizotinib inhibited P-gp, OCT1, and OCT2 in vitro at clinically relevant concentrations. Use caution with co-administration of P-gp, OCT1, and OCT2 substrates.

#### 5.1.9 Side Effects

Rev. 8/15

See Section 3.3 for side effects.

#### 6. Translational Studies

Please refer to the MATCH Master Protocol for information on the Translational Studies.

#### 7. References

- 1. Kwak EL, Bang Y-J, Camidge DR, et al. Anaplastic Lymphoma Kinase Inhibition in Non–Small-Cell Lung Cancer. New England Journal of Medicine 2010;363:1693-703.
- 2. Camidge DR, Bang Y-J, Kwak EL, et al. Activity and safety of crizotinib in patients with ALK-positive non-small-cell lung cancer: updated results from a phase 1 study. The Lancet Oncology 2012;13:1011-9.
- 3. Shaw AT, Kim D-W, Nakagawa K, et al. Crizotinib versus Chemotherapy in Advanced ALK-Positive Lung Cancer. New England Journal of Medicine 2013;368:2385-94.
- Shaw AT, Ou S-HI, Bang Y-J, et al. Crizotinib in ROS1-Rearranged Non–Small-Cell Lung Cancer. New England Journal of Medicine 2014;DOI: 10.1056/NEJMoa1406766:null.
- Lovly CM, Gupta A, Lipson D, et al. Inflammatory myofibroblastic tumors harbor multiple potentially actionable kinase fusions. Cancer Discovery 2014;8:889-95.
- 6. Li C, Alvey C, Bello A, Wilner K, Tan W. Pharmacokinetics (PK) of crizotinib (PF-02341066) in patients with advanced non-small cell lung cancer (NSCLC) and other solid tumors. J Clin Oncol 2011;29.
- 7. Kwak E, Camidge D, Clark J, et al. Clinical activity observed in a phase I dose escalation trial of an oral c-met and ALK inhibitor, PF-02341066. J Clin Oncol 2009;27:(suppl; abstr 3509).
- 8. Weickhardt AJ, Doebele RC, Purcell WT, et al. Symptomatic reduction in free testosterone levels secondary to crizotinib use in male cancer patients. Cancer 2013:119:2383-90.
- 9. Huber KVM, Salah E, Radic B, et al. Stereospecific targeting of MTH1 by (S)-crizotinib as an anticancer strategy. Nature 2014;508:222-7.
- Shaw A, Camidge D, Engleman J, et al. Clinical activity of crizotinib in advanced non-small cell lung cancer (NSCLC) harboring ROS1 gene rearrangement. J Clin Oncol 2012.
- 11. Bergethon K, Shaw AT, Ignatius Ou S-H, et al. ROS1 Rearrangements Define a Unique Molecular Class of Lung Cancers. Journal of Clinical Oncology 2012;30:863-70.
- 12. McDermott U, Iafrate AJ, Gray NS, et al. Genomic Alterations of Anaplastic Lymphoma Kinase May Sensitize Tumors to Anaplastic Lymphoma Kinase Inhibitors. Cancer Research 2008;68:3389-95.
- 13. Yasuda H, Figueiredo-Pontes Ld, Kobayashi S, Costa D. Preclinical Rationale for Use of the Clinically Available Multitargeted Tyrosine Kinase Inhibitor Crizotinib in ROS1-Translocated Lung Cancer. Journal of Thoracic Oncology 2012;7:1086-90.
- 14. Rimkunas V, Crosby K, Kelly M, et al. Frequencies of ALK and ROS in NSCLC FFPE tumor samples utilizing a highly specific immunohistochemistry-based assay and FISH analysis. J Clin Oncol 2010;28:suppl; abstr 10536.

- 15. Cilloni D, Carturan S, Bracco E, et al. Aberrant activation of ROS1 represents a new molecular defect in chronic myelomonocytic leukemia. Leukemia Research 2013;37:520-30.
- 16. Lee J, Lee SE, Kang SY, et al. Identification of ROS1 rearrangement in gastric adenocarcinoma. Cancer 2013;119:1627-35.
- 17. Davies KD, Doebele RC. Molecular Pathways: ROS1 Fusion Proteins in Cancer. Clinical Cancer Research 2013;19:4040-5.
- 18. Weickhardt A, Nguyen T, Paskulin D, et al. ALK and ROS1 gene rearrangements detected in colorectal cancer (CRC) by fluorescence in situ hybridization (FISH). J Clin Oncol 2013;31.

### Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol G: Criztonib

#### Appendix I

Rev. 3/17 Pill Calendar

**Storage:** Store at Room Temperature

#### Rev. 12/16 Pill Calendar Directions

- 1. Take your scheduled dose of each capsule.
- 2. Any missed dose may be taken up to 6 hours prior to the next scheduled dose, otherwise it should be skipped and dosing resumed with subsequent doses.
- 3. Please bring the empty bottle or any leftover capsules and your pill calendar to your next clinic visit.
- 4. Swallow capsules whole (do not crush, dissolve, or open capsules).
- 5. Take with or without food. Taking with food may decrease nausea.

#### **Patient Pill Calendar**

This is a calendar on which you are to record the time and number of capsules you take each day. You should take your scheduled dose of each capsule. **Note the times and the number of capsules that you take each day.** If you develop any side effects, please record them and anything you would like to tell the doctor in the space provided. Bring any unused capsules and your completed pill calendar to your doctor's visits.

#### Crizotinib

| | | Date | | Time ca | apsules<br>ken | | ber of<br>es taken | Use the space below to make notes about things you would like to tell the doctor (including unusual symptoms you experience, other medicine you have taken and anything else |
|---|---|---|---|---|---|---|---|---|
| DAY | Month | Day | Year | AM | PM | AM | РМ | you think would be of interest.) |
| 1 | | | | | | | | |
| 2 | | | | | | | | |
| 3 | | | | | | | | |
| 4 | | | | | | | | |
| 5 | | | | | | | | |
| 6 | | | | | | | | |
| 7 | | | | | | | | |
| 8 | | | | | | | | |
| 9 | | | | | | | | |
| 10 | | | | | | | | |
| 11 | | | | | | | | |
| 12 | | | | | | | | |
| 13 | | | | | | | | |
| 14 | | | | | | | | |
| 15 | | | | | | | | |
| 16 | | | | | | | | |
| 17 | | | | | | | | |
| 18 | | | | | | | | |
| 19 | | | | | | | | |
| 20 | | | | | | | | |
| 21 | | | | | | | | |
| 22 | | | | | | | | |
| 23 | | | | | | | | |
| 24 | | | | | | | | |
| 25 | | | | | | | | |
| 26 | | | | | | | | |
| 27 | | | | | | | | |
| 28 | | | | | | | | |

| Patient Signature: | Date: |
|--------------------|-------|

### Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol G: Criztonib

#### Appendix II

#### CYP3A4 Inducers and Inhibitors

Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as Facts and Comparisons or Lexicomp; medical reference texts such as the Physicians' Desk Reference may also provide this information. The Principal Investigator should be alerted if the subject is taking any agent on these lists.

#### **List of CYP3A4 Inducing Agents:**

Carbamazepine Phenytoin Primidone Dexamethasone Ethosuximide Progesterone Rifabutin Glucocorticoids Rifampin Griseofulvin Modafinil Rifapentine Rofecoxib Naficillin Nelfinavir St. John's Wort Nevirapine Sulfadimidine Oxcarbazepine Sulfinpyrazone Phenobarbitol **Tipranavir** Phenylbutazone Troglitazone

#### **List of CYP3A4 Inhibitors:**

Amiodarone Mifepristone Cimetidine Nefazodone Ciprofloxacin Nelfinavir Clarithromycin Norfloxacin Delavirdine Norfluoxetine Diethyl-dithiocarbamate Ritonavir Diltiazem Roxithromycin Erythromycin Saguinavir Fluconazole Troleandomycin Fluvoxamine Voriconazole Gestodene Warfarin Grapefruit or Grapefruit juice **Amprenavir** Indanvir Atazanavir Itraconazole Miconazole Ketoconazole Telithromycin Mibefradil Verapamil

### Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol G: Criztonib

Rev. 12/16 Rev.Add13

#### Appendix III

#### **Information On Possible Drug Interactions**

### Information on Possible Interactions with Other Agents for Patients and Their Caregivers and Non-Study Healthcare Team

The patient \_\_\_\_\_ is enrolled on a clinical trial using the experimental agents **Crizotinib**. This clinical trial is sponsored by the National Cancer Institute. This form is addressed to the patient, but includes important information for others who care for this patient.

Crizotinib interacts with many drugs that are processed by your liver. Because of this, it is very important to tell your study doctors about all of your medicine before you start this study. It is also very important to tell them if you stop taking any regular medicine, or if you start taking a new medicine while you take part in this study. When you talk about your medicine with your study doctor, include medicine you buy without a prescription at the drug store (over-the-counter remedy), or herbal supplements such as St. John's wort.

Many health care prescribers can write prescriptions. You must also tell your other prescribers (doctors, physicians' assistants or nurse practitioners) that you are taking part in a clinical trial. **Bring this paper with you and keep the attached information card in your wallet**. These are the things that you and they need to know:

Crizotinib interacts with certain specific enzymes in your liver.

- The enzymes in question are CYP 2B6 and 3A4 enzymes. Crizotinib blood levels are
  affected (could be lower or higher) by some of these enzymes and taking crizotinib with
  some medicines can raise or lower the levels of crizotinib or other medicines you take (drugdrug interaction). Crizotinib must be used very carefully with other medicines that need
  these liver enzymes to be effective or to be cleared from your system.
- Other medicines may also affect the activity of the enzymes.
  - Substances that increase the enzyme's activity ("inducers") could reduce the
    effectiveness of the drug, while substances that decrease the enzyme's activity
    ("inhibitors") could result in high levels of the active drug, increasing the chance of
    harmful side effects.
    - Crizotinib should not be taken with any other drugs that are strong inducers or inhibitors of CYP 3A4. Prohibited medications include azole antifungals, some antiepileptic drugs, some antibiotics and some immunosuppressants as well as over the counter drugs such as St. John's Wort. Please check with the study investigator before prescribing or dispensing strong inhibitors/inducers of CYP 3A4. Grapefruit or grapefruit juice should also be avoided.
  - Crizotinib is considered an inhibitor of CYP 2B6 and 3A4, meaning that it can increase
    the levels of drugs that are substrates of CYP 2B6 or 3A4 with a narrow therapeurtic
    index. This can lead to harmful side effects of those medications. Avoid using or
    prescribing drugs that could be affected including but not limited to alfentanil,
    cyclosporine, dihydroergotamine, ergotamine, fentanyl, pimozide, quinidine, sirolimus,
    tacrolimus.

- Crizotinib inhibits the transport proteins P-glycoprotein, OCT1 or OCT2. Medications that are substrates for these transport proteins must be used with caution.
- You and healthcare providers who prescribe drugs for you must be careful about adding or removing any drug in this category.
- Before you start the study, your study doctor will work with your regular prescriber to switch
  any prohibited medicines that are considered "strong inducers/inhibitors or substrates of
  CYP 2B6 or 3A4."
- Your prescribers should look at a frequently-updated drug reference to see if any medicine they want to prescribe is on a list of drugs to avoid.
- Please be very careful! Over-the-counter drugs have a brand name on the label—it's
  usually big and catches your eye. They also have a generic name—it's usually small and
  located above or below the brand name, and printed in the ingredient list. Find the generic
  name and determine, with the pharmacist's help, whether there could be an adverse
  interaction.
- Be careful:
  - If you take acetaminophen regularly: You should not take more than 3 grams (six 500 mg pills, or nine 325 mg pills) a day if you are an adult or 2.4 grams (four 500 mg pills, or seven 325 mg pills) a day if you are older than 65 years of age. Read labels carefully! Acetaminophen is an ingredient in many medicines for pain, flu, and cold.
  - If you take herbal medicine regularly: You should not take St. John's wort while you are taking crizotinib.
  - Avoid consumption of grapefruit, grapefruit juice, and Seville oranges.
  - Avoid antacids and tell your doctor if you are taking any medicine for heartburn symptoms.
    - Other medicines can be a problem with your study drugs.
- You should check with your doctor or pharmacist whenever you need to use an over-thecounter medicine or herbal supplement.
- Your regular prescriber should check a medical reference or call your study doctor before prescribing any new medicine for you.

Crizotinib may interact with other drugs which can cause side effects. For this reason, it is very important to tell your study doctors of any medicines you are taking before you enroll onto this clinical trial. It is also very important to tell your doctors if you stop taking any regular medicines, or if you start taking a new medicine while you take part in this study. When you talk about your current medications with your doctors, include medicine you buy without a prescription (over-the-counter remedy), or any herbal supplements such as St. John's Wort. It is helpful to bring your medication bottles or an updated medication list with you.

| Your study doctor's name is |
|-----------------------------------|
| and he or she can be contacted at |

### INFORMATION ON POSSIBLE DRUG INTERACTIONS

You are enrolled on a clinical trial using the experimental agent **crizotinib.** This clinical trial is sponsored by the NCI. Crizotinib interacts with drugs that are processed by your liver. Because of this, it is very important to:

- ➤ Tell your doctors if you stop taking regular medicine or if you start taking a new medicine.
- ➤ Tell all of your prescribers (doctor, physicians' assistant, nurse practitioner, pharmacist) that you are taking part in a clinical trial.
- Check with your doctor or pharmacist whenever you need to use an over-the-counter medicine or herbal supplement.
- ➤ Crizotinib interacts with specific liver enzymes called CYP 2B6 and 3A4, and must be used very carefully with other medicines that interact with these enzymes.

- Before you start the study, your study doctor will work with your regular prescriber to switch any prohibited medicines that are considered "strong inducers/inhibitors or major substrates of CYP 2B6 or 3A4 with a narrow therapeutic index" or will use caution when combining Crizotinib with medications that are substrates of the transporters P-glycoprotein, OCT1 or OCT2.
- Avoid consumption of grapefruit, grapefruit juice or Seville oranges while taking crizotinib.
- ➤ Before prescribing new medicines, your regular prescribers should check a frequently-updated drug resource for a list of drugs to avoid, or contact your study doctor.

| and can be contacted at |
|-------------------------|

> Your study doctor's name is

### Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol G: Criztonib

Rev. 5/16 Appendix IV

Rev. Add13

#### **Actionable Mutations for Sub-Protocol EAY131-G**

Other novel ROS1 fusions not listed in the below table but identified by one of the designated outside laboratories as described in the MATCH Master Protocol will also be considered actionable mutations (aMOIs) at Level of Evidence Code 3. Please refer to Section 1.4.2 of the MATCH Master Protocol for more information.

| Gene | Variant ID | Variant Description | Level of Evidence |
|---|---|---|---|
| ROS1 | TMEM106B-ROS1.T3R35 | Fusion | 1 |
| ROS1 | SDC4-ROS1.S4R34.COSF1280 | Fusion | 1 |
| ROS1 | SDC4-ROS1.S2R32.COSF1265 | Fusion | 1 |
| ROS1 | YWHAE-ROS1.Y4R36 | Fusion | 1 |
| ROS1 | MSN-ROS1.M9R34 | Fusion | 1 |
| ROS1 | CEP85L-ROS1.C8R36 | Fusion | 1 |
| ROS1 | CCDC6-ROS1.C5R35.1 | Fusion | 1 |
| ROS1 | KDELR2-ROS1.K5Rintron34 | Fusion | 1 |
| ROS1 | KDELR2-ROS1.K5R35 | Fusion | 1 |
| ROS1 | PWWP2A-ROS1.P1R36 | Fusion | 1 |
| ROS1 | SDC4-ROS1.S2R34 | Fusion | 1 |
| ROS1 | HLA_A-ROS1.H7R34 | Fusion | 1 |
| ROS1 | SLC34A2-<br>ROS1.S4R34.COSF1198 | Fusion | 1 |
| ROS1 | GOPC-ROS1.G8R35.COSF1139 | Fusion | 1 |
| ROS1 | EZR-ROS1.E10R35 | Fusion | 1 |
| ROS1 | SDC4-ROS1.S4R32.COSF1278 | Fusion | 1 |
| ROS1 | KIAA1598-ROS1.K11R36 | Fusion | 1 |
| ROS1 | CLIP1-ROS1.C19R36 | Fusion | 1 |
| ROS1 | CD74-ROS1.C6R34.COSF1200 | Fusion | 1 |
| ROS1 | PPFIBP1-ROS1.P9R35 | Fusion | 1 |
| ROS1 | LRIG3-ROS1.L16R35.COSF1269 | Fusion | 1 |
| ROS1 | TPM3-ROS1.T3R36 | Fusion | 1 |
| ROS1 | NFKB2-ROS1.N13R36 | Fusion | 1 |
| ROS1 | SLC34A2-<br>ROS1.S13R34.COSF1261 | Fusion | 1 |
| ROS1 | CD74-ROS1.C6R35.COSF1478 | Fusion | 1 |

| Gene | Variant ID | Variant Description | Level of Evidence |
|---|---|---|---|
| ROS1 | SLC34A2-ROS1.S13R36 | Fusion | 1 |
| ROS1 | ZCCHC8-ROS1.Z2R36 | Fusion | 1 |
| ROS1 | CD74-ROS1.C6R32.COSF1202 | Fusion | 1 |
| ROS1 | CD74-ROS1.C4R33.NGS | Fusion | 1 |
| ROS1 | ERC1-ROS1.E11R36 | Fusion | 1 |
| ROS1 | SLC34A2-<br>ROS1.S13R32.COSF1259 | Fusion | 1 |
| ROS1 | TPM3-ROS1.T7R35.COSF1273 | Fusion | 1 |
| ROS1 | TFG-ROS1.T4R35 | Fusion | 1 |
| ROS1 | EZR-ROS1.E10R34.COSF1267 | Fusion | 1 |
| ROS1 | SLC34A2-<br>ROS1.S4R32.COSF1196 | Fusion | 1 |
| ROS1 | NCOR2-ROS1.N7R36 | Fusion | 1 |
| ROS1 | MYO5A-ROS1.M23R35 | Fusion | 1 |
| ROS1 | GOPC-ROS1.G4R36.COSF1188 | Fusion | 1 |

## Molecular Analysis for Therapy Choice (MATCH) MATCH Treatment Subprotocol G: Criztonib

#### Appendix V

### **Medications That May Cause QTc Prolongation**

| During that are generally | Drugs that in some reports have been <u>associated</u> with Torsades | Drugs that, in some reports, have been weakly associated with Torsades de Pointes and/or QTc prolongation but that are unlikely to be a risk for |
|---|---|---|
| Drugs that are generally accepted to have a risk of causing Torsades de Pointes | de Pointes and/or QTc prolongation but at this time lack substantial evidence for causing Torsades de Pointes | Torsades de Pointes when used in usual recommended dosages and in subjects without other risk factors (e.g., concomitant QTc prolonging drugs, bradycardia, electrolyte disturbances, |
| | Torsades de Pointes | congenital long QTc syndrome, concomitant drugs that inhibit metabolism) |
| Generic/Brand Name | Generic/Brand Name | Generic/Brand Name |
| Amiodarone /Cordarone® | Alfuzosin /Uroxatral® | Amitriptyline /Elavil® |
| Amiodarone /Pacerone® | Amantadine /Symmetrel® | Ciprofloxacin /Cipro® |
| Arsenic trioxide<br>/Trisenox® | Atazanavir /Reyataz® | Citalopram /Celexa® |
| Astemizole /Hismanal® | Azithromycin /Zithromax® | Clomipramine /Anafranil® |
| Bepridil /Vascor® | Chloral hydrate /Noctec® | Desipramine /Pertofrane® |
| Chloroquine /Aralen® | Clozapine /Clozaril® | Diphenhydramine /Benadryl® |
| Chlorpromazine<br>/Thorazine® | Dolasetron /Anzemet® | Diphenhydramine /Nytol® |
| Cisapride /Propulsid® | Dronedarone /Multaq® | Doxepin /Sinequan® |
| Clarithromycin /Biaxin® | Felbamate /Felbatrol® | Fluconazole /Diflucan® |
| Disopyramide /Norpace® | Flecainide /Tambocor® | Fluoxetine /Sarafem® |
| Dofetilide /Tikosyn® | Foscarnet /Foscavir® | Fluoxetine /Prozac® |
| Domperidone /Motilium® | Fosphenytoin /Cerebyx® | Galantamine /Reminyl® |
| Droperidol /Inapsine® | Gatifloxacin /Tequin® | Imipramine /Norfranil® |
| Erythromycin /Erythrocin® | Gemifloxacin /Factive® | Itraconazole /Sporanox® |
| Erythromycin /E.E.S.® | Granisetron /Kytril® | Ketoconazole /Nizoral® |
| Halofantrine /Halfan® | Indapamide /Lozol® | Mexiletine /Mexitil® |
| Haloperidol /Haldol® | Isradipine /Dynacirc® | Nortriptyline /Pamelor® |
| Ibutilide /Corvert® | Lapatinib /Tykerb® | Paroxetine /Paxil® |
| Levomethadyl /Orlaam® | Lapatinib /Tyverb® | Protriptyline /Vivactil® |
| Mesoridazine /Serentil® | Levofloxacin /Levaquin® | Sertraline /Zoloft® |
| Methadone /Dolophine® | Lithium /Lithobid® | Solifenacin /VESIcare® |
| Methadone /Methadose® | Lithium /Eskalith® | Trimethoprim-Sulfa /Sulfa® |
| Pentamidine /Pentam® | Moexipril/HCTZ /Uniretic® | Trimethoprim-Sulfa /Bactrim® |
| Pentamidine /NebuPent® | Moxifloxacin /Avelox® | Trimipramine /Surmontil® |
| Pimozide /Orap® | Nicardipine /Cardene® | |
| Probucol /Lorelco® | Nilotinib /Tasigna® | |

| Drugs that are generally accepted to have a risk of causing Torsades de Pointes | Drugs that in some reports have been <u>associated</u> with Torsades de Pointes and/or QTc prolongation but at this time lack substantial evidence for causing Torsades de Pointes | Drugs that, in some reports, have been weakly associated with Torsades de Pointes and/or QTc prolongation but that are unlikely to be a risk for Torsades de Pointes when used in usual recommended dosages and in subjects without other risk factors (e.g., concomitant QTc prolonging drugs, bradycardia, electrolyte disturbances, congenital long QTc syndrome, concomitant drugs that inhibit metabolism) |
|---|---|---|
| Generic/Brand Name | Generic/Brand Name | Generic/Brand Name |
| Procainamide /Pronestyl® | Octreotide /Sandostatin® | |
| Procainamide /Procan® | Ofloxacin /Floxin® | |
| Quinidine /Cardioquin® | Ondansetron /Zofran® | |
| Quinidine /Quinaglute® | Oxytocin /Pitocin® | |
| Sotalol /Betapace® | Paliperidone /Invega® | |
| Sparfloxacin /Zagam® | Perflutren lipid microspheres /Definity® | |
| Terfenadine /Seldane® | Quetiapine /Seroquel® | |
| Thioridazine /Mellaril® | Ranolazine /Ranexa® | |
| | Risperidone /Risperdal® | |
| | Roxithromycin* /Rulide® | |
| | Sertindole /Serlect® | |
| | Sertindole /Serdolect® | |
| | Sunitinib /Sutent® | |
| | Tacrolimus /Prograf® | |
| | Tamoxifen /Nolvadex® | |
| | Telithromycin /Ketek® | |
| | Tizanidine /Zanaflex® | |
| | Vardenafil /Levitra® | |
| | Venlafaxine /Effexor® | |
| | Voriconazole /VFend® | |
| | Ziprasidone /Geodon® | |